CLINICAL TRIAL: NCT00148031
Title: Improving Hepatitis C Treatment in Injection Drug Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Steven Batki, M.D., Prinicpal Investigator, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNY UMU IRB # 4929; R01DA016764 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C; Liver Diseases; Drug Abuse; Alcoholism
Keywords: behavior modification; health care service utilization; hepatitis C,; injection drug use; therapy compliance; alcoholism; alcohol abuse; prevention; drug abuse; liver disorder; HCV; methadone
MeSH Terms: conditions — Hepatitis C; Liver Diseases; Substance-Related Disorders; Alcoholism; Patient Acceptance of Health Care; Patient Compliance; Digestive System Diseases | interventions — Ribavirin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): On-site (MMT Clinic) HCV evaluation and treatment
  Interventions: Drug: Pegylated Interferon and Ribavirin; Behavioral: Psychosocial; Behavioral: On-site (MMT Clinic) HCV evaluation and treatment
- 2 (Active Comparator): Off-site (GI Clinic) HCV evaluation and treatment
  Interventions: Drug: Pegylated Interferon and Ribavirin; Behavioral: Psychosocial; Behavioral: Off-site HCV evaluation and treatment

INTERVENTIONS:
Drug: Pegylated Interferon and Ribavirin — Both groups with receive the same medical intervention but offered at different locations
Behavioral: Psychosocial — Assessment of the likelihood of HCV treatment initiation and completion
Behavioral: On-site (MMT Clinic) HCV evaluation and treatment — Standard HCV treatment with Pegylated Interferon and Ribavirin
  Arms: 1
Behavioral: Off-site HCV evaluation and treatment — Standard HCV treatment with Pegylated Interferon and Ribavirin
  Arms: 2

SUMMARY:
The overall goal of the research project is to improve the outcome of medical care for injection drug users (IDUs) with Hepatitis C viral (HCV) infection.

Hypothesis: An intervention designed to improve the rate of HCV treatment completion and sustained virologic response (SVR) in IDUs will increase access by integrating HCV medical care into a substance abuse treatment program.

DETAILED DESCRIPTION:
The overall goal of the proposed health services research project is to improve the outcome of medical care for injection drug users (IDUs) with Hepatitis C viral (HCV) infection. This will be done by testing an intervention designed to improve the rate of HCV treatment completion and sustained virologic response (SVR) in IDUs. This intervention will increase access by integrating HCV medical care into a substance abuse treatment program. HCV infection is endemic among IDUs, and is associated with significant medical morbidity. While antiviral treatments are improving rapidly, providing HCV medical care for IDUs remains problematic for a number of reasons. IDUs often do not have adequate access to HCV diagnosis and treatment services, and they may have co-morbid psychiatric diagnoses that affect the ability to withstand the demands of HCV treatment. Therefore, this study will also examine psychiatric disorders and psychiatric symptoms in IDUs who are infected with Hepatitis C virus.

The proposed project is a five-year program consisting of a controlled clinical trial, studying 220 patients with HCV infection enrolled in methadone maintenance treatment (MMT). The HCV Medical Care Study is a randomized trial to test the efficacy of On-site HCV Medical Care provided at the MMT program versus Off-site care at the Gastroenterology (GI) Clinic. HCV antibody positive MMT patients (N=220) will be randomly assigned to receive HCV medical services either through an integrated delivery model located on-site in the MMT clinic, or through usual off-site referral to the GI Clinic. The main outcomes will be the rates of attaining SVR and completion of HCV treatment, as well as other measures of HCV-related health outcomes and quality of life. Participants will be evaluated for Axis I psychiatric diagnoses and will complete psychiatric measures at monthly intervals throughout the study. Psychiatric diagnosis will be made using the Structured Psychiatric Interview for the DSM-IV (SCID) and psychiatric symptom severity will be assessed for depression, mania, anxiety, and psychosis. Drug use measures, and quality of life measures will also be obtained. These data are expected to yield new knowledge about the efficacy of providing on-site HVC medical care in substance abuse treatment programs. They will provide a comparison of psychiatric diagnoses and psychiatric symptom presentation in HCV positive IDUs who choose to receive HCV treatment and those who do not choose to follow through with HCV treatment and will describe changes in psychiatric symptoms before, during, and after HCV medical care. Finally, the studies will also provide information about the influence of psychiatric symptoms and drug and alcohol use on HCV medical outcomes such as treatment completion and SVR.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age.
2. Enrolled in outpatient methadone maintenance treatment for greater than 3 months.
3. Hepatitis C RNA positive.
4. Willingness to accept HCV treatment.
5. Subject has non-VA (Veteran's Administration) medical insurance or is willing to bear any and all expenses associated with Hepatitis C medical treatment.

Exclusion Criteria:

1. In need of inpatient drug or alcohol detoxification.
2. Currently receiving the standard Hepatitis C treatment
3. Unable to give adequate informed consent.
4. Pregnant, nursing, or planning to become pregnant during HCV treatment or within 6 months following completion of treatment.
5. Male subject who has a female sexual partner who is pregnant or planning to become pregnant at any time during HCV treatment or within 6 months following completion of treatment.
6. Female subject or male subject who has a female sexual partner who is of child bearing years and not using two medically approved forms of contraception.
7. Subject has made a commitment to attend residential care psychiatric or drug/alcohol rehabilitation, which would lead to unavailability to attend regularly scheduled medical care and research visits.
8. Subject did not attend all required screening appointments.
9. Subject has a legal proceeding whose outcome may lead to incarceration within 3 months of intake.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2003-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of On-site versus Off-site delivery of HCV medical care for methadone maintenance treatment (MMT) patients, as evaluated by the proportion of patients achieving sustained virological response (SVR). | 5 years

SECONDARY OUTCOMES:
psychiatric diagnoses and symptom severity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Batki, MD, Principal Investigator — State University of New York, Upstate Medical University - Department of Psychiatry
Locations (2):
- United States (2):
  - Crouse Chemical Dependency Treatment Services, Syracuse, New York
  - SUNY Upstate Medical University - Department of Gastroenterology, Syracuse, New York

REFERENCES:
- [Background] Cornell, M.E., Peek, R.M.H., Batki, S.L. (2002) Hepatitis C in an Upstate New York methadone treatment population: Preliminary analysis. Drug and Alcohol Dependence 66:S36-37.
- [Background] Batki, S.L., Srinath, A.K., Cornell, M.E., Bowman, M., Peek, R.M.H., Wade, M., Dimmock, J., Abdul-Hamid, M. (2005) Depression and Substance Use in Methadone Patients with Hepatitis C. American Journal on Addictions 14:304-5.
- [Result] Batki, S.L., Canfield, K.M., Cole, C., Smyth, E., Pham, H., Ploutz-Snyder, R.; Amodio, K., Manser, K., Knoeller, G., Strutynski, K., Levine, R., Dimmock J.A. (2007) (abstract) Psychiatric diagnosis and psychiatric symptom severity in methadone treatment patients with untreated hepatitis C virus infection. American Journal on Addictions, 16:316-17.
- [Result] Batki, S.L., Canfield, K., Lundell, S., Levine, R., Donohue, L., Amodio, K. (oral presentation) Characteristics of opioid-dependent patients seeking Hepatitis C treatment. College on the Problems of Drug Dependence, Orlando, June.
- [Result] Batki, S.L., Canfield, K.M., Cole, C., Ploutz-Snyder, R., Dimmock, J., Pham, H., Smythe, E. (oral presentation) Quality of life in MMT patients with untreated HCV infection. College on the Problems of Drug Dependence, Scottsdale, June 2006.
- [Result] Batki, S.L.; Canfield, K.; Cole, C.; Smyth, E.; Ploutz-Snyder, R.; Levine, R.; Amodio, K.; Knoeller, G.; Strutynski, K.; Manser, K.; Dimmock, J.A. (oral presentation) Hepatitis C treatment progress by methadone maintenance patients: Preliminary analysis of a trial of co-located treatment. College on the Problems of Drug Dependence, Quebec City, June 2007
- [Result] Batki, S.L., Canfield, K.M., Smyth, E., Amodio, K., Manser, K., Levine, R.A. (poster presentation) Effects of medical and psychiatric comorbidity on HCV treatment eligibility in methadone maintenance. College on the Problems of Drug Dependence, Annual Meeting, San Juan, Puerto Rico June, 2008
- See also: State University of New York, Upstate Medical University — http://www.upstate.edu